CLINICAL TRIAL: NCT00166855
Title: Clinical Implication of Bone Marrow Perfusion Patterns Imaged by Dynamic MRI in Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9361701200
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-05

CONDITIONS: Multiple Myeloma, Newly Diagnosed
Keywords: angiogenesis; bone marrow perfusion; dynamic MRI; multiple myeloma; prognosis
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Procedure: dynamic MRI and bone marrow sampling

SUMMARY:
Background: Multiple myeloma (MM) is a clonal plasma cell neoplasm characterized by proliferation of neoplastic plasma cells in bone marrow (BM). So far, it is an incurable disease and the median survival time of MM patients is only three to four years. Till now, whether the extent of angiogenesis in BM of MM patients serves as an important and independent prognostic factor is still debated. In this study, we would like to have the BM perfusion status imaged by dynamic MRI to mimic the macroscopic vascular densities of BM, and thereafter, the BM perfusion status, the clinical outcome of the MM patients, and the angiogenesis related biological markers will be correlated.

Methods: About 35 to 50 MM patients, included newly diagnosed patients or the patients who will undertake the special treatment, are enrolled in this study. The thoraco-lumbar spine is scanned by the MRI, and the BM perfusion status is obtained by contrast-enhanced dynamic MRI. Meanwhile, the patients undertake BM biopsy at one site or two sites and the BM aspirates are also obtained and separated into BM plasma and BM mononuclear cells (BMMC) by Ficoll-Hypaque centrifugation. The angiogenesis related genes expression profiles of the BMMC will be determined by cDNA microarrays and some of them, like VEGF, bFGF, and PDGF, will be semiquantified by real-time PCR. The levels of related proteins will be determined by ELISA. The BM plasma samples are further applied to proteomic analysis to screen the novel molecules with clinical relevance.

Prospects: BM perfusion patterns imaged by dynamic MRI can predict the clinical outcome of MM, and are correlated with the angiogenesis relevant biological markers in BM.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a clonal plasma cell neoplasm characterized by proliferation of abnormal plasma cells in bone marrow (BM) that secrete a monoclonal paraprotein (M-protein) in serum and/or urine, and by osteolytic bone destructions. So far, it is an incurable disease and its pathogenesis is largely unknown. The median survival time of MM patients is only three to four years, and then the patients will die on either the disease or its complications [Barlogie et al, 2004].

There are several independent prognostic factors for MM, like high levels of beta-2 microglobulin, hypodiploidy chromosome content, deletion of chromosome 13q14 and also the extent of angiogenesis, shown by microvascular density (MVD), in BM [Fonseca et al, 2004; Kumar et al, 2002; Pruneri et al, 2002; Sezer et al, 2000]. It has been suggested that MM progressed from an avascular to a vascular phase (active MM) accompanied by a significant increase in MVD in BM [Rajkumar et al, 2002], which is promoted by the angiogenesis related factors, like VEGF, bFGF, and PDGF, which were performed like a paracrine or autocrine loops secreted by MM cells per se or the adjacent BM stromal cells [Gupta et al, 2001; Kumar et al, 2003; Ria et al, 2003; Vacca et al, 2003]. It has been reported that higher MVD in BM at the time of initial diagnosis was associated with shorter OS and PFS in patients undergoing autologous transplantation for MM than the patients with lower MVD [Kumar et al, 2004]. Those angiogenesis related factors may provide disease monitoring but also a potent novel therapeutic approach to over come resistance to therapies and thereby improve patient outcome [Podar et al, 2004]. Interestingly, the patients with deletion of chromosome 13q14 have higher MVD in BM than the patients without [Schreiber 2000], which hinted that the grave prognosis of deletion of chromosome 13q14 might be a result of dysregulation of angiogenesis in BM. However, on the other hand, absence of clinical prognostic value of VEGF and MVD in MM had also been reported by other investigators [Ahn et al, 2001; Choi et al, 2002]. In MM, whether the MVD in BM and the related biological markers, like VEGF, bFGF, and PDGF can serve as prognostic factors are still debate [Rajkumar et al, 2001; Vacca et al, 2001]. There are possible two reasons for the debate, the first one is that the distribution of neoplastic foci within the BM of MM are not homogenous, therefore the microvascular densities calculated from a single site BM specimen are hard to represent the total angiogenesis within the BM; the second one is that the angiogenesis related biological markers, such as VEGF, bFGF, and PDGF, in MM are largely studied on the plasmas obtained from peripheral blood rather than BM, and this is a critical issue for the cytokines secreted from either MM cells or adjacent stromal cells are mostly paracrines or autocrines and the levels of VEGF, bFGF, PDGF are higher in BM than in peripheral blood [Di Raimondo et al, 2000].

Reviewing the literature, dynamic contrast-enhanced MRI has been used to evaluate the potential of vertebral fractures in MM [Scherer et al, 2002a & 2002b], to quantify significant changes of BM microcirculation during conventional treatment [Rahmouni et al, 1993] or treatment with thalidomide combined with chemotherapy [Wasser et al, 2004], which may be a novel and non-invasive tool to approach the clinical outcomes of MM patients [Moehler et al, 2001]. In short, MR imaging of the spine was performed with a 1.5-T superconducting system (Magnetom Vision Plus; Siemens, Erlangen, Germany). A phase-array spine-coil was used, and a routine fast spin-echo T1-weighted sequence (repletion time msec/echo time msec, 600/12; turbo factor of three; section thickness, 4 mm; field of view, 28cm) was performed in the midsagittal plane and covered the area from T11 through the sacrum. A dynamic contrast-enhanced MR study was then performed (section thickness, 10 mm; field of view, 28 cm) at the midsection of the vertebral body and covered the same area. The pulse sequence used was a turbo fast low-grade shot gradient-echo sequence (8.5/4.0; prepulse inversion time, 160 msec; flip angle, 10°; acquisition matrix, 72x128). Acquisition time was 0.89 second with 0.11-second delay. In total, 100 dynamic images were obtained within 100 seconds (one frame per second) in each subject. After the initial 100-second scanning, the scanning were prolong to 600 seconds with the scan rate 1 frame per 10 seconds (1 seconds scan and 9 seconds delay). An injection of 0.1 mmol per kilogram of body weight gadopentetate dimeglumine (Magnevist; Schering, Berlin, Germany) was administrated by the power injector through a 21-gauge intravenous catheter that was inserted in the right antecubital vein previously. A brief constant injection rate of 2.0ml/sec were used. This injection was immediately followed with a 20-ml saline flush at the same injection rate. Dynamic imaging started when the injection of the contrast material commenced.

Signal intensity values were measured in an operator-defined region of interests (ROIs). The musculoskeletal radiologist (T.T.F.S., with 15 years experience) places the ROIs were placed with the aid of a cursor and a graphic display device, along the border of high-signal-intensity bone marrow on T1 weighted images covered the entire bone marrow of each vertebra. One vertebral body was covered by one ROI measurement. The ROI was measured separately for each of selected lumbar vertebrae (L2, L3 and L4) in each subject. The signal intensity values derived from the ROI measured in each vertebral body were then plotted against time to obtain a time-signal intensity curve (Fig 1) for each vertebral body. The baseline value for signal intensity (SIbase) on a time- signal intensity curve was defined as the mean signal intensity from the first three images. The maximum signal intensity (SImax) was defined as the maximum value of the first rapidly rising part of the time-signal intensity curve. The time to peak contrast enhancement was defined as the time (Trise) between SIbase and SImax. After the peak, which usually occurred about 40 seconds after the start of injection, the time-signal intensity curve entered an equilibrium phase that lasted about 30 seconds. The total 100-second imaging time encompassed both the first rapid rise in the curve and the early equilibrium phase. In our study, the SIbase and SImax were measured only from the first rapidly rising curve. For the semiquantitative analysis, the peak enhancement ratio peak was calculated for each ROI as (SImax - SIbase)/SIbase and average enhancement slope (average slope) was defined as (SImax - SIbase)/ Trise for each ROI. The initial slope was measured as the most steep uprising slope from the early rapid-rising part of time intensity curve. The mean value was calculated from the parameters of the L3, L3 and L4 vertebrae and represented for each subject. In our preliminary study, like others [Moehler et al, 2001], this constructed images performed by dynamic contrast-enhanced MRI, which mimic the perfusion status within bone marrow, had been correlated with distinct clinical outcomes in our acute myeloid leukemia and MM patients in a preliminary study.

Accordingly, we would like to have the BM perfusion status imaged by dynamic MRI to mimic the macroscopic vascular densities of BM, and thereafter, the BM perfusion status, the clinical outcome of the MM patients, and the angiogenesis related biological markers will be correlated.

ELIGIBILITY:
Inclusion Criteria:multiple myeloma, newly diagnosed -

Exclusion Criteria:nil, except for the patients disagree MRI study nor bone marrow sampling

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-07; Study Completion 2009-07

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Yi Huang, M.D., Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan